CLINICAL TRIAL: NCT01585688
Title: A Phase I/II Study of Immunotherapy With hLL1-DOX in Patients With Non-Hodgkin's Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL)
Brief Title: Phase I/II Study of hLL1-DOX in Relapsed NHL and CLL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to lack of efficacy, as a result, the stability program for the drug product was discontinued
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hLL1-DOX-02
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2020-02

CONDITIONS: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia
Keywords: NHL; CLL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — milatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hLL1-DOX (Experimental)
  Interventions: Drug: hLL1-DOX (IMMU-115)

INTERVENTIONS:
Drug: hLL1-DOX (IMMU-115) — hLL1-DOX is administered intravenously at one of 4 dose levels on days 1, 4, 8 and 11 of 21-day treatment cycles, with up to 8 cycles administered.
  Other Names: IMMU-115

SUMMARY:
The primary objectives are to evaluate the safety and tolerability of hLL1-DOX, and to determine the maximum tolerated dose (MTD) regimen (in terms of a dose and its associated dosing schedule). The secondary objectives are to obtain information on efficacy, pharmacodynamics, pharmacokinetics, and immunogenicity, and to determine the optimal dose for subsequent studies.

DETAILED DESCRIPTION:
Patients receive hLL1-DOX at one of 4 dose levels administered on Days 1, 4, 8 and 11 of 21-day treatment cycles which are continued in the absence of progression or unacceptable toxicity up to a total of 8 cycles. After treatment, follow-up will be done at 4, 8 and 12 weeks post-treatment and will continue to be done every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years
* Able to provide signed, informed consent
* Histologically confirmed diagnosis of recurrent B-cell non-Hodgkin's lymphoma (any histology by WHO criteria) or recurrent chronic lymphocytic leukemia (by NCI criteria) (Reference Appendix C)
* Received at least one prior treatment with standard therapy (previous antibody therapy is acceptable)
* Measurable disease at least one lesion ≥ 1.5 cm for NHL and ALC > 5,000 for CLL
* Adequate performance status (≥ 70 Karnofsky scale) with an estimated life expectancy of at least 6 months

  --Documented negative hepatitis B screen, per NCCN guidelines (hepatitis B surface antigen/antibodies, core antigen/antibodies, hepatitis B e-antigen)
* At least 12 weeks beyond stem cell transplant and 4 weeks beyond chemotherapy or immunotherapy, major surgery, other experimental treatments, or radiation therapy to the index lesions, and with all acute toxicities from prior therapy resolved to less than Grade 2 toxicity by NCI CTC version 4.0
* Laboratory parameters:

Adequate hematology without ongoing transfusional support Hemoglobin >/= 10 g/dL Absolute neutrophil count >/= 1.5 x 10 9/L Platelets >/= 75 x 10 9/L Creatinine and bilirubin </= 1.5 x IULN AST and ALT </= 2.5 x IULN

-Adequate cardiac function (MUGA scan or 2-D ECHO with LVEF ≥ 55%, EKG with no medically relevant arrhythmia uncontrolled on medications)

Exclusion Criteria:

* -Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study until at least 12 weeks after the last milatuzumab infusion
* Prior therapy with other human or humanized monoclonal antibodies, unless HAHA tested and negative
* Prior treatment with trastuzumab
* Bulky disease by CT, defined as any single mass > 10 cm in its greatest diameter
* Known HIV positive or active hepatitis B or C, or presence of hepatitis B surface antigens or presence of hepatitis C antibody
* New York Heart Classification III or IV heart disease (see Appendix G). Other severe cardiovascular or cardiopulmonary disease, including COPD
* Baseline BNP > 2 x IULN
* Patients with uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities will be excluded
* Patients with recent (≤ 6 months) cardiac angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias will be excluded
* Known autoimmune disease or presence of autoimmune phenomena
* At least 7 days beyond any infection requiring intravenous antibiotic use (Oral antibiotics may be administered prophylactically as clinically indicated)
* Systemic corticosteroids within 2 weeks, except low dose regimens (prednisone, ≤ 20 mg/day, or equivalent) which may continue if unchanged
* Substance abuse or other concurrent medical or psychiatric conditions that, in the Investigator's opinion, could confound study interpretation or affect the patient's ability to tolerate or complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of hLL1-DOX | These assessments will be done routinely during treatment & changes at 4, 8 & 12 weeks after treatment
  NCI CTCAE version 4.0 is used to grade all adverse events
All patients who were treated and meet the efficacy criteria for response assessment will be included in the analysis of efficacy | During treatment and the changes at 4, 8 and 12 weeks after treatment and then every 3 months for up to 2 years
  For the primary efficacy evaluations, the proportion of responders (defined as patients with a best response of PR or CR) will be tabulated for each dose level. In addition, the progression-free survival (PFS, as measured from start of treatment to disease progression, death or last follow-up) will be summarized using Kaplan-Meier survival analysis methods.
  Similarly, for responders at each dose level, the duration of response (DR, as measured from time of first response to relapse or last follow-up) will also be summarized using Kaplan- Meier survival analysis methods, if appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Pius P Maliakal, PhD, Study Director — Gilead Sciences; Francois Wilhelm, MD,PhD, Study Chair — Gilead Sciences
Locations (6):
- United States (6):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - IU Health Goshen Center for Cancer Care, Goshen, Indiana
  - UMass Memorial Cancer Center of Excellence, Worcester, Massachusetts
  - John Theurer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - U.T. MD Anderson Cancer Center Houston, Houston, Texas